CLINICAL TRIAL: NCT01560351
Title: Repeated Low-frequency Transcranial Magnetic Stimulation Reduces Cue-induced Craving: a Randomized, Prospective, Double-blind, Sham-controlled, Cross-over Study
Acronym: STIMJEU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BRD/11/6-M
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Pathological Gambling
Keywords: Pathological gambling; craving; repeated Transcranial Magnetic Stimulation; craving cues
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS (Experimental): Session of repeated low-frequency Transcranial Magnetic Stimulation
  Interventions: Device: rTMS
- Placebo (Sham Comparator): Sessions of sham rTMS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Two sessions of repeated Transcranial Magnetic Stimulation (real rTMS and sham rTMS) are planned for each participant, at interval of 4 weeks, in a random order.

SUMMARY:
The aim of this study is to evaluate the effect of repeated low-frequency Transcranial Magnetic Stimulation (rTMS) of the right dorsolateral prefrontal cortex, combined with gambling cues, on gambling craving. Participants are pathological gamblers. A single real stimulation and a single shame stimulation are administered in a random order for each participant (cross-over study).

ELIGIBILITY:
Inclusion criteria:

* Pathological gambler (DSM-IV criteria)
* Seeking treatment at the University Hospital of Nantes
* Right-handed
* 18-65 years old
* Increase in the intensity (at least 50%) of the gambling craving with gambling cues

Non-inclusion criteria:

* pregnant woman
* no effective contraception
* Substance use disorders (excluding nicotine)
* Benzodiazepine use
* Chronic neurological disease
* History of head injury
* History of neurosurgery
* Cochlear implant or other metal objects in the head
* History of Transcranial Magnetic Stimulation or repeated Transcranial
* Magnetic Stimulation
* Difficult to read or write French

Exclusion criteria:

* Occurrence of side effects (like seizures)
* Psychoactive substance use 12 hours before the rTMS (excluding nicotine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS)
  Cue-induced craving is evaluated using a VAS, immediately before and immediately after the administration of the craving cues, and immediately after the rTMS session (real and sham).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS)
  Cue-induced craving kinetics : cue-induced craving is evaluated using a VAS every 5 minutes until its intensity returns to baseline.
Gambling Craving Scale (GACS)
  Cue-induced craving is also evaluated using the GACS, immediately before and immediately after the administration of the craving cues, immediately after the rTMS session, and every 5 minutes until its intensity returns to baseline.
blood pressure
  Cue-induced craving is also evaluated using the measure of the blood pressure, immediately before and immediately after the administration of the craving cues, immediately after the rTMS session, and every 5 minutes until its intensity returns to baseline.
heart rate
  Cue-induced craving is also evaluated using the measure of the heart rate, immediately before and immediately after the administration of the craving cues, immediately after the rTMS session, and every 5 minutes until its intensity returns to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anne SAUVAGET, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes, Nantes, France

REFERENCES:
- See also: Click here for more information about this study and about excessive gambling — http://www.crje.fr